CLINICAL TRIAL: NCT04130295
Title: Influence of Wearable Intensive Nerve Stimulation on Spasticity and Function in Persons With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 787
Record Dates: First submitted 2019-10-07; First posted 2019-10-17 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injuries; Spasticity, Muscle
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wearable intensive nerve stimulation (Experimental): The device will be worn on the upper calf with each session of stimulation lasting 60 minutes after which the device will turn off for 60 minutes before turning back on. Participants will be instructed to wear the device for 5 hours a day in order to receive three one our sessions of stimulation.
  Interventions: Other: Wearable intensive nerve stimulator

INTERVENTIONS:
Other: Wearable intensive nerve stimulator — The wearable device consists of 2 leads that provide biphasic, with alternating lead phase, asymmetrical rectangular current at a pulse duration of 0.28 msec, a randomly varying pulse frequency between 60-100 Hz, with a maximum intensity of 100mA.

SUMMARY:
Spasticity is muscle spasms, bouncing (clonus) or stiffness that can negatively impact the quality of life of people with spinal cord injury (SCI). In people with spinal cord injury, spasticity can limit muscle control of the arms and hands and cause pain, discomfort, and frustration. Transcutaneous electrical stimulation has been shown to reduce spasticity after SCI. However, this type of stimulation's effects during prolonged, at-home use has not been well studied. Additionally, traditional stimulation techniques are often only available in the clinic. Therefore, this study aims to identify if wearable intensive nerve stimulation decreases spasticity in the legs of people with SCI, and if this intervention is usable and desirable to individuals with SCI.

DETAILED DESCRIPTION:
Involuntary muscle activation, also referred to as spasticity is a common characteristic of spinal cord injuries. It can present as stiffness, clonus, and spasms that can impact a person's ability to perform daily tasks. Over half of individuals with spinal cord injuries that have spasticity report medication alone does not control the spasticity. Because of this clinical research is investigation different ways to manage spasticity.

Stretching and vibration have demonstrated the ability to reduce spasticity but only for short periods of time requiring repeated use of the intervention. Additionally, vibration devices are not very practical to implement at home due to their high cost. Due to these factors, a solution that could be used multiple times a day and remains cost effective is needed.

Transcutaneous electrical stimulation (TENS) has also demonstrated effectiveness in reducing spasticity after one session but shows greater benefit when it is able to be used for multiple sessions. A wearable intensive nerve stimulator (WINS) device has been shown to be safe for daily wear which makes it a feasible solution to address spasticity at home. Research has not yet looked at the efficacy of using the WINS device for spasticity and this study proposes to begin to fill that gap.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-65 years of age
* Have sustained cervical or thoracic SCI at least 6 months prior to initiating participation in study
* Any ISNCSCI severity classification (A, B, C, or D)
* Have self-reported spasticity and at the time of screening demonstrate an FSE angle of ≤ 75 degrees on the pendulum test or ≥ 4 beats of clonus on the drop test
* May participate if utilizing oral prescription medications for control of spasticity
* Ability and willingness to consent and authorize use of personal health information

Exclusion Criteria:

* Severe contractures of the leg/foot to be stimulated (decided during pre-assessment) that limit passive movement of the hip, knee, or ankle more than 50% of normal range of motion or presence of other orthopedic pathology that would adversely influence participation in the protocol
* Any implanted catheter such as but not limited to CSF shunt, baclofen pump, or the presence of a pacemaker, implanted automatic internal cardioverter defibrillator (AICD, other cardiac implants and or conditions)
* Severe pain or hypersensitivity of the leg to be stimulated (decided during pre-assessment)
* Uncontrolled edema of the leg to be stimulated (decided during pre-assessment)
* Current pregnancy
* Lumbar spinal cord injury level
* Inability or unwillingness to consent and authorize use of personal health information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Spasticity | Week 1, Week 2, Week 3, and Week 7
  Instrumented Pendulum Test: Participants will be in a semi-reclined position on a therapy mat. The examiner will then bring the participants knee into full extension before dropping the foot. The examiner will observe the number of oscillations to determine muscle stretch-induced activity
Satisfaction and Adherence Questionnaire | Week 7
  Participant will answer questions about how likely they would be to continue to use the intervention at home.
Spinal Cord Injury - Spasticity Evaluation Tool | Twice per week
  a Questionnaire used to characterize the impact of spasticity on a participant's ability to perform everyday occupations.

SECONDARY OUTCOMES:
Manual Ankle Clonus Test | Week 1, Week 2, Week 3, and Week 7
  Participants are positioned in supine with legs extended. The examine will move each foot individually into dorsiflexion and observe the number of beats of clonus. This will be used to determine muscle-stretch induced activity of the lower limb
Ankle Drop Test | Week 1, Week 2, Week 3, and Week 7
  Participants are seated on the edge of the table with one leg fully extended. The examiner holds the test leg 10 cm above a wooden block before dropping it onot the block to observe the duration of clonus if there is any. The test will determine muscle-stretch induced activity.
Flexor Spasms | Week 1, Week 2, Week 3, and Week 7
  Participants are in supine with the hip and knee extended. The examiner will then stimulate the foot with a safety pin and observe movement of the great toe, ankle dorsiflexion, and hip and knee flexion. This tool is used to determine spasticity
Instrumented Flexor Reflex Response | Week 1, Week 2, Week 3, and Week 7
  Participants will be positioned in supine with knee and hip extended. The examiner will stimulate the foot with an electrical stimulus and observe movement of the great toe, ankle dorsiflexion, and hip and knee flexion. The tool is used to determine spasticity in the lower limb.
Global Impression of Change Scale | Week 1, Week 2, Week 3, and Week 7
  a self-report measure designed to quantify the participant's improvement or deterioration over time. This tool will be used to rate how spasticity is impacting the participant's function. The scale is an 11 point scale from -5, representing that spasticity is much worse, to 5, which reports that spasticity is much better. Participants will use this scale to evaluate spasticity at the ankle, hip, and knee.
Adherence Data | Week 3, Week 4, Week 5, and Week 7
  Adherence data will be collected from the device, which stores data on duration and number of therapy sessions completed each day. This tool will be used to measure participant adherence.
Assessing neurophysiological aspects of spasticity | Week 1, Week 2, Week 3, and Week 7
  Electrodes will be placed on the quadriceps, hamstring, tibialis anterior, and soleus muscles to observe muscle activity during rest and testing. Biomechanical measurements of lower extremity movement will be made using inertial motion capture equipment (Xsens)

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States